CLINICAL TRIAL: NCT04949698
Title: "Risk Factors for Pregnancy-related Thrombotic Microangiopathies Retrospective Study of the Effect of Plasma Exchange on Prognosis of Pregnancy-related Thrombotic Microangiopathies"
Brief Title: Risk Factors and the Effect of Plasma Exchange on Prognosis of Pregnancy-related Thrombotic Microangiopathies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020304
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy-related Thrombotic Microangiopathies
Keywords: pregnancy; thrombotic microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — Plasma Exchange

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No TMA: parturients without thrombotic microangiopathies
  Interventions: Device: plasma exchange
- TMA with plasma exchange: parturients with thrombotic microangiopathies, and treated with plasma exchange
  Interventions: Device: plasma exchange
- TMA without plasma exchange: parturients with thrombotic microangiopathies, but not treated with plasma exchange
  Interventions: Device: plasma exchange

INTERVENTIONS:
Device: plasma exchange — Plasma exchange was performed daily for five times or until platelet level returned to normal

SUMMARY:
Early identification of the risk factors of pregnancy-related thrombotic microangiopathies can help us reduce the complications of such patients and increase the survival rate of patients. In addition, it is still controversial whether patients with pregnancy-related thrombotic microvessels should receive plasma therapy.

DETAILED DESCRIPTION:
"Objective: To evaluate the risk factors of pregnancy-related thrombotic microangiopathies and the effect of plasma exchange on the prognosis (recovery status of renal function, recovery status of platelets, survival or death within 28 days).

Design: A retrospective analysis of pregnant patients admitted to the ICU from 2015 to 2019. According to the outcome indicator of the occurrence of pregnancy-related thrombotic microangiopathies, they were divided into thrombotic microangiopathies group and non-thrombotic microangiopathies group. Patients in the pregnancy-related thrombotic microangiopathy group were divided into plasma exchange combined non-plasma exchange group according to whether they received plasma exchange. Collect the clinical data of the patients, and analyze the data using SPSS 1 7.0 statistical software package. The measurement data were compared by paired t test and one-way analysis of variance; the count data were compared by χ2 test. Compare the differences of the indicators between the two groups and analyze the risk factors of pregnancy-related thrombotic microangiopathies. Then compare whether there is a difference in the prognosis between the plasma exchange group and the non-plasma exchange group."

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients admitted to the Department of critical care medicine, the Third Hospital of Peking University from 2015 to 2019

Exclusion Criteria:

* NO

Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study is for puerpera with or without TMA, so patients should be female only
Study Population: Pregnant patients admitted to the Department of critical care medicine, the Third Hospital of Peking University from 2015 to 2019
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
TMA happen | 28th day after ICU admission
  pregnancy associated thrombotic microangiopathy happen or not at 28th day after ICU admission

SECONDARY OUTCOMES:
renal function | 28th day after ICU admission
  renal function at 28th day after ICU admission
platelet level | 28th day after ICU admission
  platelet level at 28th day after ICU admission
survival rate | 28th day after ICU admission
  survival rate at 28th day after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Min Yi, chief physician, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Undecided